CLINICAL TRIAL: NCT07227155
Title: Hematopoietic Cell Transplant and Gene Therapy for Non-Malignant Blood Disorders Biobank Resource (BMT CTN 2402)
Brief Title: The HOPE Biobank Resource (BMT CTN 2402 HOPE)
Acronym: HOPE Resource
Status: Not yet recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BMT CTN 2402
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Aplastic Anemias; Hemoglobinopathies; Bone Marrow Failure
Keywords: Biorepository; Biospecimens; Allogenic Transplant; Gene Therapy
MeSH Terms: conditions — Anemia, Aplastic; Hemoglobinopathies; Bone Marrow Failure Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, germline (skin, hair, nails), bone marrow, stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, multicenter study that will establish a repository of biospecimens and clinical data from patients undergoing hematopoietic stem cell transplant (HCT) or gene therapy (GT) for treatment of non-malignant blood diseases.

DETAILED DESCRIPTION:
This is a prospective, multicenter, study that will establish a repository of biospecimens and clinical data from patients undergoing hematopoietic stem cell transplant (HCT) or gene therapy (GT) for treatment of non-malignant blood diseases. The enrollment goal is 375 participants and up to all consenting 100 related donors (approximately 100 are anticipated), accrued over 4 years. Participants will be followed until the end of study, but continued collection of specimens and clinical data may continue to allow up to 15 years of follow-up for all enrolled participants if funds are available. Participants with a diagnosis of Aplastic Anemia or Hemoglobinopathies or bone marrow failure undergoing HCT or GT for management of their underlying disease. There is no treatment intervention in this study. Treatment will be at the provider's discretion. Participants will provide blood and other biospecimens pre and post-intervention at specified intervals. 375 participants and approximately 100 related donors will be enrolled from 35 sites.

ELIGIBILITY:
HCT/GT Inclusion:

1. Patients with a diagnosis of Aplastic Anemia (AA), hemoglobinopathies or bone marrow failure from other causes except for malignant diseases will be eligible for enrollment on this protocol:

   1. AA will be defined as having peripheral blood cytopenias with a hypocellular bone marrow for age and a clinical diagnosis of aplastic anemia as determined by their treating physicians.
   2. Hemoglobinopathies include sickle cell disease or thalassemia. Patients receiving potentially curative therapy with HCT or GT for hemoglobinopathies will be eligible for this study.
   3. Individuals with bone marrow failure due to clinical or molecularly diagnosed inherited bone marrow failure, inborn errors of immunity or other cause will be included.
2. Patients must receive an HCT or GT for management of their underlying disease. Allogeneic transplants including all conditioning regimens, donors, and GVHD prophylaxis regimens are eligible. This study does not define how the transplant or transplant-supportive care will be performed.
3. Patients or their legal guardian must consent to participate in the CIBMTR "Protocol for a Research Database for Hematopoietic Cell Transplantation and Marrow Toxic Injuries" (NCT 1166009) to allow linkage with the longitudinal clinical data collected by CIBMTR.
4. All ages minorities, sexes and genders are eligible for the study, but participants must weigh at least 10 kilograms (kg) at the time of study enrollment given the volume and number of blood draws required.
5. All participants or parent/legal guardian must sign an informed consent for this study. If there are questions regarding a patient's eligibility for the study, contact the Protocol Team for review and discussion by emailing bmtctn2402@emmes.com.

HCT/GT Exclusion

1. Patients with aplastic anemia or hemoglobinopathies who are not pursuing allogeneic HCT or GT.
2. Active malignancy.
3. Hematologic malignancy or therapy for a prior hematologic malignancy in the previous five 5 years.
4. Weight ≤ 10.0 kg at time of study enrollment.
5. Prior autologous or allogeneic transplant.

Related Donor Inclusion:

1. All related donors for eligible recipients undergoing allogeneic HCT for AA, hemoglobinopathies, or bone marrow failure as defined in the recipient eligibility criteria above are eligible. Note: HCT recipient participants will remain eligible if the related donor declines to participate in the study.

Related Donor Exclusion:

1. Donor weight ≤ 10.0 kg at time of study enrollment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing HCT or GT for treatment of Non-malignant blood disorders: Aplastic Anemia, Hemoglobinopathies or Bone Marrow Failure. Related donors of enrolled participants undergoing HCT are also eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2026-03-27 (Estimated); Primary Completion 2031-03-30 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
Develop a biorepository that will establish mechanistic insights and biologic correlates to key casues of fialure of HCT and GT for Non-malignant Diseases (NMD). | 5 Years
  Retention of biospecimen samples with DNA
Identify new therapeutic targets for NMD and HCT or GT related complications leading to development of more targeted and effective therapies. | 5 Years
  Retention of biospecimen samples with DNA

IPD SHARING:
Plan to Share IPD: Undecided